CLINICAL TRIAL: NCT03918070
Title: Multicenter Observatory to Assess the Yukon Choice PC & the Yukon Chrome PC Sirolimus Eluting Bioabsorbable Polymer Stents Systems in Routine Clinical Practice
Brief Title: Observatory to Assess the Yukon Choice PC & the Yukon Chrome PC Sirolimus Eluting Bioabsorbable Polymer Stents Systems
Acronym: YuChooSeR
Status: Active, not recruiting | Type: Observational
Sponsor: Translumina GmbH (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A03455-50
Record Dates: First submitted 2019-04-12; First posted 2019-04-17 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Coronaropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Yukon Choice PC and Yukon Chrome PC — The Yukon Choice PC & the Yukon Chrome PC Sirolimus Eluting Bioabsorbable Polymer Coronary Stent Systems are indicated for improving coronary luminal diameter in patients with symptomatic ischemic heart disease.

SUMMARY:
The TRANSLUMINA GmbH YuChooSeR Observatory is a prospective, multicentric post-marketing observatory designed to evaluate large scale safety and reliability of the Yukon Choice PC and the Yukon Chrome PC stents systems use in routine, clinical practice.

This based observatory will enroll 3000 patients to 30 sites in France.

DETAILED DESCRIPTION:
TRANSLUMINA GmbH has launched clinical programs to demonstrate the safety and efficacy of its technology.

The Translumina Yukon Choice PC drug-eluting stent, coated with Rapamycin (Sirolimus) and the biodegradable component polylactide (PLA), has an excellent history of pre-clinical and clinical results.

The Yukon Chrome PC has the identical coating technique and coating properties (dosage, thickness) like the clinically proven Yukon Choice PC.

In two independent trials ISAR-TEST 3 and ISAR-TEST 4 the Yukon DES platform showed angiographic and clinical equivalence with the Cypher stent after 1 year and 3 years of follow-up.

Latest clinical data, published by G.Stefanini et al, show the excellent long-term outcome of the Yukon biodegradable polymer DES technology in a meta-analysis, comparing the clinical outcome after 4 years in more than 4000 patients with the Cypher stent. This analysis shows for the first time that the definite Very Late Stent Thrombosis (VLST) can be reduced statistically significant by using the biodegradable PLA polymer coating technology of the Yukon DES.

An additional sub-group analysis shows also benefit in difficult patient groups like diabetics and patients with acute myocardial infarkt.

Due to this excellent clinical outcome the Yukon DES technology is recommended by the latest ESC guidelines for myocardial revascularization.

The final 5 years long-term clinical follow-up of the ISAR-TEST 4 randomized controlled clinical trial showed excellent safety and efficacy data for the Yukon DES when compared with the Cypher and Xience V stent. The definite and probable stent thrombosis was only 1,2% for the Yukon compared to 1,4% and 2,4% for the 2 permanent polymer coated competitor DES.

In a continued approach to collect safety and efficiency data on its products, TRANSLUMINA GmbH is determined to collect safety and efficiency information at a very large scale. Based on all this, the Yukon Choice PC & the Yukon Chrome PC stents have been designed to treat coronary arteries in a relatively easy and simple-to-achieve manner, while providing a higher level of clinical efficacy.

Additionally, the Observatory is aimed to provide a learning tool that will help to define best practices/techniques as all results will be fed back to participants and to a larger audience through publications.

In this Observatory, analyses will be performed per clinical presentation and per stent type.

ELIGIBILITY:
Inclusion Criteria:

* Any patient suitable for implantation with a Yukon Choice PC or a Yukon Chrome PC stent according to current guidelines can be enrolled in this observatory
* Patient must be over 18 years old.

Exclusion Criteria:

* Patient not able to understand the information given for collection, transfer and processing of personal data before participation, may not be enrolled in this observatory.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic ischemic heart disease requiring stenting. All patients selected by the investigator to receive a Yukon Choice PC and/or a Yukon Chrome PC stent can be enrolled. Patient must be over 18 years old and be informed verbally and in writing about the nature and aim of the study.
Sampling Method: Non-Probability Sample
Enrollment: 2722 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-05-24 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is Target Lesion Failure (TLF) rate at 12 months follow-up | 12 months follow-up
  Target Lesion Failure (TLF) is defined as the composite of cardiac death, target-vessel myocardial Infarction and clinically indicated target lesion revascularization (TLR) by percutaneous or surgical methods.

SECONDARY OUTCOMES:
Device Success | 12 months follow-up
  Device Success defined as successful delivery and deployment of the assigned device at the intended target lesion and successful withdrawal of the delivery system with attainment of final in-stent residual stenosis of <30% (by visual estimation)
Procedure Success | 12 months follow-up
  Procedure Success defined as Device Success without the occurrence of ischemia-driven major adverse cardiac event (ID-MACE) during the hospital stay to a maximum of first seven days post index procedure.
Reperfusion | 12 months follow-up
  Reperfusion measured by TIMI flow at the end of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Didié Tchétché, Dr, Principal Investigator — Clinique Pasteur
Locations (19):
- France (19):
  - Clinique Axium, Aix-en-Provence
  - Hopital A. Schweitzer - Ghca, Colmar
  - Centre Hospitalier de Compiègnes, Compiègne
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Clinique Louis Pasteur, Essey-lès-Nancy
  - GHM Grenoble, Grenoble
  - Centre Hospitalier Haguenau, Haguenau
  - Hopital privé Beauregard, Marseille
  - Clinique Pont de Chaume, Montauban
  - Hopital Privé du Confluent, Nantes
  - Centre Hospitalier de Périgueux, Périgueux
  - Centre Hospitalier de Quimper, Quimper
  - Clinique Saint Hilaire, Rennes
  - Polyclinique Saint-Laurent, Rennes
  - Centre Hospitalier de Soissons, Soissons
  - Centre Hospitalier de Saint Malo, St-Malo
  - Centre Hospitalier de Bigorre, Tarbes
  - Clinique Pasteur, Toulouse
  - Centre Hospitalier de Vannes, Vannes

IPD SHARING:
Plan to Share IPD: No